CLINICAL TRIAL: NCT04904380
Title: Impact of Simulation-enhanced Peer Learning With Novel Tools on Maternal and Newborn Mortality Plus Knowledge, Skills Retention and Decision Making by Front-line Health Workers in Southwestern Uganda
Brief Title: Impact of New Tools of Simulation-enhanced Peer Learning on Neonatal and Maternal Mortality
Acronym: Sim-II
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mbarara University of Science and Technology (Other)
Collaborators: University of Calgary (Other); The ELMA Foundation (Other); Alberta Children's Hospital Research Institute (Other); Laerdal Foundation (Other); International Development Research Centre, Canada (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2020/MUST-5/SIM-II
Record Dates: First submitted 2021-04-30; First posted 2021-05-27 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-04

CONDITIONS: Neonatal Mortality; Maternal Mortality
MeSH Terms: conditions — Maternal Death | interventions — Hemoglobin, Sickle; Air

STUDY DESIGN:
Intervention Model Description: Randomized cluster trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): HMS, HBS and peer learning in combination with AIR and PRISMS
  Interventions: Other: Active peer learning
- Comparison arm (Active Comparator): HMS, HBS and peer learning in combination with PRISMS but no AIR
  Interventions: Other: Active peer learning

INTERVENTIONS:
Other: Active peer learning — HMS, HBS and peer learning in combination with AIR and PRISMS
  Other Names: Enhanced HMS and HBS with PRISMS and AIR

SUMMARY:
In the vast majority of developing nations, frontline birth attendants are often the only care providers responsible for newborn care including newborn resuscitation, thermal care, feeding and administration of medications. These midwives need knowledge and skills to provide all these newborn clinical care needs. However, frontline birth attendants in these circumstances are seldom exposed to the training and decision support tools that would empower them to holistically assess, decide and manage newborn babies in their care. Current training opportunities are fragmented and need to be administered as a comprehensive package.

A combination approach to training, skills retention, and the use of decision support tools such as Protecting Infants Remotely by SMS (PRISMS) and Augmented Infant Resuscitator (AIR) may provide a comprehensive package for the acquisition and retention of knowledge and skills on newborn care and empower birth attendants to provide effective, timely interventions.

DETAILED DESCRIPTION:
The investigators will implement the Sim for Life Impart, Retain, Empower and Monitor (IREM) module at the University of Jos teaching Hospital and 4 high volume health facilities in Tanzania in addition to the Uganda sites. We propose to implement the program with all its components for each of the partner institutions.

The Sim for Life IREM module combines four strategies: Impart skills using Helping Babies Survive (HBS)/Helping Mothers Survive (HMS) courses, Retain skills (Simulation), Empower birth attendants (PRISMS and AIR) and Monitor progress objectively. The simulation sessions for health facilities will be conducted using the peer to peer learning methodology which equips participants with the skills to facilitate simulation scenarios in their health facilities. The scenarios will be provided by the Sim for life team. The topics for the scenarios will be based on common maternal and newborn illnesses like post-partum hemorrhage, pre-eclampsia, birth asphyxia, neonatal sepsis and prematurity.

All health facilities in this study will require smart phones for the PRISMS application, resuscitation practice tables, source of electricity to charge a phone, practice manikins / associated practice supplies and peer learning cards.

ELIGIBILITY:
Inclusion Criteria:

* Newborns babies
* Mothers delivering at participating health facilities
* Health workers providing maternal and newborn care services at participating health facilities

Exclusion Criteria:

* Health care workers not providing maternal and newborn care services
* Male patients
* Non pregnant female patients seeking care at participating health facilities

Min Age: 0 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3456 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Neonatal mortality | Neonatal mortality at 6 months
  Neonatal mortality
Neonatal mortality | Neonatal mortality at 18 months
  Neonatal mortality
Maternal mortality | Maternal mortality at 6 months
  Maternal mortality
Maternal mortality | Maternal mortality at 18 months
  Maternal mortality

SECONDARY OUTCOMES:
Length of stay in hospital | 18 months
  Number of days as length of stay
Completeness of newborn assessment | At admission
  Completeness of newborn assessment checklist

CONTACTS AND LOCATIONS:
Overall Officials: Data Santorino, MD, Principal Investigator — Mbarara University of Science and Technology

IPD SHARING:
Plan to Share IPD: No
Data includes sensitive material with video records